CLINICAL TRIAL: NCT02600481
Title: Comparison of the Impacts of Prolonged Low-pressure and Standard-pressure Pneumoperitoneum on Myocardial and Pulmonary Injuries After Robot-assisted Surgery in the Trendelenburg Position: a Bi-center, Randomized Controlled Trial
Brief Title: Impacts of Different Pressure Pneumoperitoneum on Myocardial and Pulmonary Injuries After Robot-assisted Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huadong Hospital (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015K060
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Prostatic Neoplasms; Urinary Bladder Neoplasms
Keywords: standard-pressure pneumoperitoneum; prolonged pneumoperitoneum; myocardial injuries; troponin T(TnT); Trendelenburg position; chest CT scan; low-pressure pneumoperitoneum; robot-assisted surgery
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- low-pressure pneumoperitoneum group (Experimental): Subjects assigned to the low-pressure pneumoperitoneum group will receive 7-10 mm Hg carbon dioxide pneumoperitoneum, and the expected duration is longer than 3 hours to complete robot-assisted surgeries in the Trendelenburg position;
  Interventions: Procedure: low-pressure pneumoperitoneum
- standard-pressure pneumoperitoneum group (Active Comparator): Subjects assigned to the standard-pressure pneumoperitoneum group will receive 12-16 mm Hg carbon dioxide pneumoperitoneum, which is expected lasted longer than 3 hours to complete robot-assisted surgeries in the Trendelenburg position;
  Interventions: Procedure: standard-pressure pneumoperitoneum

INTERVENTIONS:
Procedure: low-pressure pneumoperitoneum — Using low-pressure(between 7-10 mm Hg ) pneumoperitoneum to complete robot-assisted surgeries,such as radical prostatectomy or cystectomy.
  Arms: low-pressure pneumoperitoneum group
Procedure: standard-pressure pneumoperitoneum — Using standard-pressure (between 12-16 mm Hg )pneumoperitoneum to complete robot-assisted surgeries,such as radical prostatectomy or cystectomy.
  Arms: standard-pressure pneumoperitoneum group

SUMMARY:
This study is aimed to determine whether low- and standard-pressure pneumoperitoneum have different impacts on troponin T（TnT) level as well as pulmonary complications after prolonged robot-assisted surgeries in the Trendelenburg position.

DETAILED DESCRIPTION:
The hypothesis of this study is based on several studies reported that increased postoperative troponin T(TnT) level was significantly associated with 30-day mortality, and some other reports showed that low-pressure pneumoperitoneum had better haemodynamic outcome than that of standard-pressure pneumoperitoneum. Hence, we hypothesize that different pneumoperitoneal pressure may lead to different levels of TnT after prolonged robot-assisted surgeries.

This clinical trial will be conducted in Huadong Hospital Affiliated to Fudan University and Ruijin Hospital Shanghai Jiao Tong University School of Medicine,both are tertiary hospitals in Shanghai, China.

After signing the Informed Consent, subjects who meet the eligibility criteria will be randomly assigned to low- or standard-pressure pneumoperitoneum group.The randomization plans will be implemented using statistical software R, and will be stored in an online database.These subjects will be recruited from January 1st 2016 to December 31st 2017.

TnT is set as the primary endpoint for this trial to evaluate the myocardial injuries, and will be measured for each patient who will undergo in-patient robot-assisted urological surgery within 24 hours postoperatively using the fourth-generation high-sensitivity TnT assay.

The total sample size will be 280.With 140 patients in each of the two treatment groups, the power will be at least 0.70 to detect an increment of TnT level among 80% of subjects.Chest CT scan is used to diagnose the pulmonary complications on the third day postoperatively.

Data will be collected to analysize whether prolonged different intraperitoneal pressure has different impacts on cardiopulmonary injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo Robot-assisted radical prostatectomy or other robot-assisted urological surgeries last longer than 3 hours
* Patients who are classified as American Society of Anesthesiologists（ASA）I and II
* Patient's preoperative troponin T(TnT) level is normal

Exclusion Criteria:

* Patients with preoperative cardiopulmonary dysfunction who can not understand prolonged surgeries in the Trendelenburg position：severe pulmonary dysfunction or New York Heart Association(NYHA) classification is Ⅲ-Ⅳ.
* Body Mass Index>30.
* Any intraoperative situation as follows：1. Any cause to cancel operation or change robot-assisted surgery to open surgery 2. Intraoperative cardiovascular accidents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Troponin T level is set as the marker of myocardial injuries after robot-assisted surgeries | Within the first 24 hours after prolonged robot-assisted surgeries

SECONDARY OUTCOMES:
Chest CT scan is used to determine pulmonary complications | On the third day after prolonged robot-assisted surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Gu, Doctor, Study Chair — Huadong Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Finkelstein J, Eckersberger E, Sadri H, Taneja SS, Lepor H, Djavan B. Open Versus Laparoscopic Versus Robot-Assisted Laparoscopic Prostatectomy: The European and US Experience. Rev Urol. 2010 Winter;12(1):35-43. PMID 20428292
- [Background] Orvieto MA, Patel VR. Evolution of robot-assisted radical prostatectomy. Scand J Surg. 2009;98(2):76-88. doi: 10.1177/145749690909800203. PMID 19799045
- [Background] Hakimi AA, Feder M, Ghavamian R. Minimally invasive approaches to prostate cancer: a review of the current literature. Urol J. 2007 Summer;4(3):130-7. PMID 17987573
- [Background] Meininger D, Byhahn C, Bueck M, Binder J, Kramer W, Kessler P, Westphal K. Effects of prolonged pneumoperitoneum on hemodynamics and acid-base balance during totally endoscopic robot-assisted radical prostatectomies. World J Surg. 2002 Dec;26(12):1423-7. doi: 10.1007/s00268-002-6404-7. Epub 2002 Sep 26. PMID 12297911
- [Background] Yiannakopoulou ECh, Nikiteas N, Perrea D, Tsigris C. Effect of laparoscopic surgery on oxidative stress response: systematic review. Surg Laparosc Endosc Percutan Tech. 2013 Apr;23(2):101-8. doi: 10.1097/SLE.0b013e3182827b33. PMID 23579502
- [Background] Sharma KC, Kabinoff G, Ducheine Y, Tierney J, Brandstetter RD. Laparoscopic surgery and its potential for medical complications. Heart Lung. 1997 Jan-Feb;26(1):52-64; quiz 65-7. doi: 10.1016/s0147-9563(97)90009-1. PMID 9013221
- [Background] Leduc LJ, Mitchell A. Intestinal ischemia after laparoscopic cholecystectomy. JSLS. 2006 Apr-Jun;10(2):236-8. PMID 16882427
- [Background] de Cleva R, Silva FP, Zilberstein B, Machado DJ. Acute renal failure due to abdominal compartment syndrome: report on four cases and literature review. Rev Hosp Clin Fac Med Sao Paulo. 2001 Jul-Aug;56(4):123-30. doi: 10.1590/s0041-87812001000400006. PMID 11717720
- [Background] Imamoglu M, Sapan L, Tekelioglu Y, Sarihan H. Long-term effects of elevated intra-abdominal pressure on testes an experimental model of laparoscopy. Urol J. 2013 Sep 26;10(3):953-9. PMID 24078502
- [Background] Joris JL, Chiche JD, Canivet JL, Jacquet NJ, Legros JJ, Lamy ML. Hemodynamic changes induced by laparoscopy and their endocrine correlates: effects of clonidine. J Am Coll Cardiol. 1998 Nov;32(5):1389-96. doi: 10.1016/s0735-1097(98)00406-9. PMID 9809953
- [Background] Russo A, Marana E, Viviani D, Polidori L, Colicci S, Mettimano M, Proietti R, Di Stasio E. Diastolic function: the influence of pneumoperitoneum and Trendelenburg positioning during laparoscopic hysterectomy. Eur J Anaesthesiol. 2009 Nov;26(11):923-7. doi: 10.1097/EJA.0b013e32832cb3c9. PMID 19696680
- [Background] Sharma KC, Brandstetter RD, Brensilver JM, Jung LD. Cardiopulmonary physiology and pathophysiology as a consequence of laparoscopic surgery. Chest. 1996 Sep;110(3):810-5. doi: 10.1378/chest.110.3.810. No abstract available. PMID 8797429
- [Background] Wahba RW, Beique F, Kleiman SJ. Cardiopulmonary function and laparoscopic cholecystectomy. Can J Anaesth. 1995 Jan;42(1):51-63. doi: 10.1007/BF03010572. PMID 7889585
- [Background] Hanaoka M, Hara Y, Fujiogi M, Fujisawa N, Kawakami M, Shioiri S, Tanaka M, Yasuno M. Pulmonary edema after laparoscopic hepatectomy in a patient with Budd-Chiari syndrome-associated hepatocellular carcinoma. Asian J Endosc Surg. 2015 May;8(2):197-200. doi: 10.1111/ases.12152. PMID 25913587
- [Background] Aydin V, Kabukcu HK, Sahin N, Mesci A, Arici AG, Kahveci G, Ozmete O. Comparison of pressure and volume-controlled ventilation in laparoscopic cholecystectomy operations. Clin Respir J. 2016 May;10(3):342-9. doi: 10.1111/crj.12223. Epub 2014 Nov 14. PMID 25307158
- [Background] Lebowitz P, Yedlin A, Hakimi AA, Bryan-Brown C, Richards M, Ghavamian R. Respiratory gas exchange during robotic-assisted laparoscopic radical prostatectomy. J Clin Anesth. 2015 Sep;27(6):470-5. doi: 10.1016/j.jclinane.2015.06.001. Epub 2015 Jul 3. PMID 26144913
- [Background] Kanwer DB, Kaman L, Nedounsejiane M, Medhi B, Verma GR, Bala I. Comparative study of low pressure versus standard pressure pneumoperitoneum in laparoscopic cholecystectomy--a randomised controlled trial. Trop Gastroenterol. 2009 Jul-Sep;30(3):171-4. PMID 20306755
- [Background] Hua J, Gong J, Yao L, Zhou B, Song Z. Low-pressure versus standard-pressure pneumoperitoneum for laparoscopic cholecystectomy: a systematic review and meta-analysis. Am J Surg. 2014 Jul;208(1):143-50. doi: 10.1016/j.amjsurg.2013.09.027. Epub 2014 Jan 16. PMID 24503370
- [Background] van Waes JA, Nathoe HM, de Graaff JC, Kemperman H, de Borst GJ, Peelen LM, van Klei WA; Cardiac Health After Surgery (CHASE) Investigators. Myocardial injury after noncardiac surgery and its association with short-term mortality. Circulation. 2013 Jun 11;127(23):2264-71. doi: 10.1161/CIRCULATIONAHA.113.002128. Epub 2013 May 10. PMID 23667270
- [Background] Ozturk TC, Unluer E, Denizbasi A, Guneysel O, Onur O. Can NT-proBNP be used as a criterion for heart failure hospitalization in emergency room? J Res Med Sci. 2011 Dec;16(12):1564-71. PMID 22973364
- [Background] Argyra E, Theodoraki K, Rellia P, Marinis A, Voros D, Polymeneas G. Atrial and brain natriuretic peptide changes in an experimental model of intra-abdominal hypertension. J Surg Res. 2013 Oct;184(2):937-43. doi: 10.1016/j.jss.2013.03.036. Epub 2013 Mar 31. PMID 23608621
- [Background] Vascular Events In Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Devereaux PJ, Chan MT, Alonso-Coello P, Walsh M, Berwanger O, Villar JC, Wang CY, Garutti RI, Jacka MJ, Sigamani A, Srinathan S, Biccard BM, Chow CK, Abraham V, Tiboni M, Pettit S, Szczeklik W, Lurati Buse G, Botto F, Guyatt G, Heels-Ansdell D, Sessler DI, Thorlund K, Garg AX, Mrkobrada M, Thomas S, Rodseth RN, Pearse RM, Thabane L, McQueen MJ, VanHelder T, Bhandari M, Bosch J, Kurz A, Polanczyk C, Malaga G, Nagele P, Le Manach Y, Leuwer M, Yusuf S. Association between postoperative troponin levels and 30-day mortality among patients undergoing noncardiac surgery. JAMA. 2012 Jun 6;307(21):2295-304. doi: 10.1001/jama.2012.5502. PMID 22706835
- [Background] Davarci I, Karcioglu M, Tuzcu K, Inanoglu K, Yetim TD, Motor S, Ulutas KT, Yuksel R. Evidence for negative effects of elevated intra-abdominal pressure on pulmonary mechanics and oxidative stress. ScientificWorldJournal. 2015;2015:612642. doi: 10.1155/2015/612642. Epub 2015 Jan 20. PMID 25685845
- [Background] Awad H, Santilli S, Ohr M, Roth A, Yan W, Fernandez S, Roth S, Patel V. The effects of steep trendelenburg positioning on intraocular pressure during robotic radical prostatectomy. Anesth Analg. 2009 Aug;109(2):473-8. doi: 10.1213/ane.0b013e3181a9098f. PMID 19608821
- [Background] Falabella A, Moore-Jeffries E, Sullivan MJ, Nelson R, Lew M. Cardiac function during steep Trendelenburg position and CO2 pneumoperitoneum for robotic-assisted prostatectomy: a trans-oesophageal Doppler probe study. Int J Med Robot. 2007 Dec;3(4):312-5. doi: 10.1002/rcs.165. PMID 18200624
- [Background] Kalmar AF, Foubert L, Hendrickx JF, Mottrie A, Absalom A, Mortier EP, Struys MM. Influence of steep Trendelenburg position and CO(2) pneumoperitoneum on cardiovascular, cerebrovascular, and respiratory homeostasis during robotic prostatectomy. Br J Anaesth. 2010 Apr;104(4):433-9. doi: 10.1093/bja/aeq018. Epub 2010 Feb 18. PMID 20167583
- [Background] Park EY, Koo BN, Min KT, Nam SH. The effect of pneumoperitoneum in the steep Trendelenburg position on cerebral oxygenation. Acta Anaesthesiol Scand. 2009 Aug;53(7):895-9. doi: 10.1111/j.1399-6576.2009.01991.x. Epub 2009 May 6. PMID 19426238
- [Derived] Zhang X, Wei J, Song X, Zhang Y, Qian W, Sheng L, Shen Z, Yang L, Dong R, Gu W. Comparison of the impact of prolonged low-pressure and standard-pressure pneumoperitoneum on myocardial injury after robot-assisted surgery in the Trendelenburg position: study protocol for a randomized controlled trial. Trials. 2016 Oct 10;17(1):488. doi: 10.1186/s13063-016-1609-5. PMID 27724965
- See also: Click here for more information about this study:the study's four objectives were to determine the diagnostic criteria, characteristics, predictors, and 30-day outcomes of MINS(myocardial injury after noncardiac surgery, MINS). — http://www.ncbi.nlm.nih.gov/pubmed/?term=24534856